CLINICAL TRIAL: NCT00172952
Title: National Taiwan University Hospital
Brief Title: The Role of SNP of ECM and MMP on the Development of Pathological High Myopia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700339
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-06

CONDITIONS: Myopia
Keywords: high myopia, genomic
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
To study the clinical characteristics and inheritance of pathological myopia in Taiwanese patients.

DETAILED DESCRIPTION:
High myopia (pathological myopia) is caused by excessive axial elongation that primarily involves the ora-equatorial area and the posterior pole. Pathological myopia often accompanied by glaucoma, cataracts, macular degeneration, and retinal detachment, leading to blindness when the damage to the retina is extremely severe. Population and family studies in Chinese have provided evidence for a geneticcomponent to pathologic myopia. Children of myopic parents are more likely to have myopia than are children of nonmyopic parents. Therefore, it is possible to search a potential candidate gene for myopia through the genomic study of pathological myopia. The retina receives the signal from the retina-RPE complexes and affects the growth of scleral coats. The changes of scleral components, collagen fibrils and proteoglycans, are noted in experimental and human myopia and induce the pathology of high myopia. It is interesting to know that individual difference of SNP in the components of scleral coat affects the response to the signal from retina-RPE complexes. The most important effectors in scleral coats are collagens, proteoglycans, MMPs and TIMPs. Therefore, the difference of SNPs in different genes might contribute the formation of scleral thinning during myopia development. In this project, we will focus on this subject by using GenomeLab SNPstream Genotyping System which is powerful and helpful for identify some specific SNPs in the regard.

ELIGIBILITY:
Inclusion Criteria:

* They are unrelated Chinese subjects with high myopia ≦-6.00D. The diagnosis of myopia is determined by the refractive error. Anisometropic individuals, with a refractive error of ≦-6.00 D for one eye and ≦-6.00 D for the other eye, with at least a 2-D difference between the two eyes, are considered unaffected

Exclusion Criteria:

* Individuals are excluded if there is known ocular disease or insult that could predispose to myopia, such as retinopathy of prematurity or early-age media opacification, or if they had a known genetic disease associated with myopia, such as Stickler or Marfan syndrome.

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600
Dates: Start 2005-06; Study Completion 2006-01

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Feng Shih, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan